CLINICAL TRIAL: NCT02160314
Title: A Clinical Study to Assess the Safety of a Disposable Intra-vaginal Device for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012119
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence, SUI, pessary
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Pessaries; Absorbent Pads

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pad (Placebo Comparator): absorbent pad control
  Interventions: Device: Absorbent pad
- pessary (Experimental): disposable, single-use pessary
  Interventions: Device: pessary

INTERVENTIONS:
Device: pessary — disposable, single-use pessary
  Arms: pessary
Device: Absorbent pad
  Other Names: placebo comparator
  Arms: pad

SUMMARY:
This study will evaluate the safety of the pessary device by objective evaluation of vaginal wall integrity and subjective assessment of comfort during in-use conditions.

ELIGIBILITY:
Inclusion Criteria:

* be female 18 years or older;
* provide written informed consent prior to study participation and been given a signed copy;
* be in generally good health as determined by the Investigator;
* have a ≥ 3 month history of experiencing Stress Urinary Incontinence (SUI) per week (self reported);
* be willing to use the pessary investigational device to control stress urinary incontinence;
* be willing to comply with study requirements and instructions;

Exclusion Criteria:

* are pregnant, lactating, or planning to become pregnant during the study;
* within 3 months post partum;
* intrauterine device (IUD) placement of less than 6 months;
* has self-reported difficulty emptying her bladder;
* a history of Toxic Shock Syndrome (TSS) or symptoms consistent with TSS;
* experience difficulty inserting or wearing an intra-vaginal device, including a tampon;
* vaginal surgery, perineal surgery, uterine surgery, or abortion (spontaneous or induced) within the past 3 months;
* has any Screening laboratory value outside the laboratory reference range considered clinically significant by the Investigator and could impact the safety of the subject or the outcome of the study; or
* for any reason, the Investigator decides that the subject should not participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Severance, MD, Principal Investigator — Radiant Research, Inc.
Locations (1):
- Study Center, Chandler, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 224 subjects signed an informed consent, 79 did not meet inclusion/exclusion criteria and were screen failed.
Groups:
- Pad Control: absorbent pad control
- Pessary: pessary: disposable, single-use
Period: Overall Study
Arm/Group | Pad Control | Pessary
Started | 73 | 72
Completed | 72 | 59
Not Completed | 1 | 13
Not completed — Adverse Event | 0 | 6
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT)
Groups:
- Pad Control: absorbent pad control
  Absorbent pad
- Total: Total of all reporting groups
Arm/Group | Pad Control | Pessary | Total
Number analyzed (Participants) | 73 | 72 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (10.24) | 53.9 (12.36) | 53.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 72 | 145
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Serious Adverse Event
Description: proportion of intent-to-treat subjects who experience a treatment-emergent serious adverse event
Time Frame: 3 month
Population: Intent-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Pad Control | Pessary
Number analyzed (Participants) | 73 | 72
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: All AEs as reported by the subject from Visit 1 (screening) through Visit 5 (exit) were recorded.
Arm/Group | Pad Control | Pessary
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 8/73 | 7/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pad Control (N=73) | Pessary (N=72)
Candida test positive (Investigations) | 4 (5) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3)
vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 4 (6) — this adverse event corresponds to vaginal spotting in 3 subjects, and vaginal bleeding in 1 subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The STUDY SITE and PRINCIPAL INVESTIGATOR agree that all data, calculations, interpretations, opinions and recommendations regarding the STUDY (hereinafter referred to as "RESULTS") shall be the property of P&G. The STUDY SITE and PRINCIPAL INVESTIGATOR agree to consider the RESULTS as INFORMATION subject to confidentiality restrictions